CLINICAL TRIAL: NCT02487212
Title: Treatment of Hypertrophic Scars Using Fractional Laser and Fractional Laser-assisted Topical Corticosteroid Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 614/2556 (EC2)
Record Dates: First submitted 2015-04-11; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hypertrophic Scars
Keywords: fractional laser; hypertrophic scar; topical corticosteroid; laser assisted delivery systems
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Clobetasol; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser+Topical corticosteroid (Active Comparator): Hypertrophic scars were treated with fractional Erbium: Yttrium aluminium garnet (YAG) (2,940-nm) laser, then 0.05% Clobetasol propionate ointment was immediately applied on the perforated scar on one side
  Interventions: Drug: 0.05% Clobetasol propionate; Device: Fractional Erbium:Yag (2,940-nm) laser
- Laser+Petrolatum gel (Placebo Comparator): Hypertrophic scars were treated with fractional Erbium: YAG (2,940-nm) laser, then topical petrolatum gel was immediately applied on the perforated scar on the other side
  Interventions: Drug: Petrolatum gel; Device: Fractional Erbium:Yag (2,940-nm) laser

INTERVENTIONS:
Drug: 0.05% Clobetasol propionate — 0.05% Clobetasol propionate was rubbed for 2 minutes on one side of the scar immediately after treated with fractional Erbium: YAG (2,940-nm) laser. The treatment was done in every 2 weeks for 4 sessions
  Arms: Laser+Topical corticosteroid
Drug: Petrolatum gel — Petrolatum gel was rubbed for 2 minutes on the other side of the scar immediately after treated with fractional Erbium: YAG (2,940-nm) laser.The treatment was done in every 2 weeks for 4 sessions
  Arms: Laser+Petrolatum gel
Device: Fractional Erbium:Yag (2,940-nm) laser — The parameter of the laser was 28 J/cm2, 5% spot density, 1 pass for the whole scar. The treatment was done in every 2 weeks for 4 sessions

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of using ablative fractional laser- assisted topical corticosteroid delivery for the treatment of hypertrophic scar.

DETAILED DESCRIPTION:
Hypertrophic scars are common conditions that cause persistent symptom and can lead to severe psychosocial impairment. Intralesional corticosteroid have been a mainstay in the treatment of hypertrophic scars. However, there are many disadvantages of corticosteroid injection such as severe pain, skin atrophy, skin thinning, steroid acne, telangiectasia and hypopigmentation.

Recent reports propose new treatment methods for hypertrophic scars with the use of fractional ablative lasers to create zones of ablation of the skin that may assisted the penetration of drugs to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with age range 18-60 years;
* Subject with hypertrophic scar from abdominal surgery for at least 3 months;
* Discontinued using oral isotretinoin for 6 months, alpha hydroxy acid or topical retinoic acid for 3 months

Exclusion Criteria:

* Subject who has skin Infection, photosensitive dermatosis or inflammatory acne on the treated area;
* Subject who smoke cigarette;
* Subject who was treated with Intralesional corticosteroid

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Scar thickness measured by digital calliper | change from baseline in scar thickness at 6 months

SECONDARY OUTCOMES:
Patient and observer scar assessment scale | Baseline, 1 month after first treatment, 1,3 and 6 months after fourth treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand